CLINICAL TRIAL: NCT05384470
Title: Detecting Drugs of Abuse Via Exhaled Breath Samples Using Differential Mobility Spectrometry
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Collaborators: VOX BIOMEDICAL LLC (Unknown)
Responsible Party: Principal Investigator, Scott Lukas, Director, McLean Imaging Center and BPRL, Mclean Hospital
Other Study IDs: 2019P001633; 5R42DA049655-04 (NIH)
Record Dates: First submitted 2022-05-16; First posted 2022-05-20 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Opiate Abuse; Marijuana Abuse; Diagnostic
Keywords: THC; marihuana; pharmacokinetics; breathalyzer
MeSH Terms: conditions — Opioid-Related Disorders; Marijuana Abuse; Disease | interventions — nabiximols

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Exhaled Breath Samples: Quantitative detection of marijuana, morphine or fentanyl through exhaled breath
  Interventions: Drug: Marihuana; Device: BID2 Instrument - breathalyzer

INTERVENTIONS:
Drug: Marihuana — Two doses of marijuana given.
Device: BID2 Instrument - breathalyzer — The commercial device that we will be testing is designed to detect breath cannabinoid concentrations utilizing Differential Mobility Spectrometry technology, and was developed by Draper, to detect a wide range of chemicals and organisms in breath. Differential Mobility Spectrometry (DMS) is a robust, data-rich, ultra-trace, chemical detection technology. Unlike gas chromatography mass spectroscopy (GCMS) systems that are large and expensive, DMS is small, portable (approximately the size of a shoe box) and is able to measure the presence of volatile organic compounds (VOC) at parts per trillion (ppt) detection levels. The participant will exhale into the device via a plastic tube and the breath sample will be analyzed in situ. The participant does not come in contact with the device itself-they will simply exhale into a tube via a disposable mouthpiece.

SUMMARY:
This Phase II STTR program consists of two major goals within the overarching goal of developing and validating a proprietary device (BID2) for marijuana and opioid detection in breath samples.

DETAILED DESCRIPTION:
This study is intended to lead to the development and demonstration of a breathalyzer instrument capable of detecting and quantitatively measuring drugs (i.e. cannabinoids and opioids) in exhaled breath (EB). Prior work on the detection of these drugs in EB by means of liquid chromatography and mass spectrometry (LC/MS) demonstrated that these compounds can be quantitatively detected, but LC/MS is slow, expensive and requires highly skilled personnel to implement. What is needed is a simple and inexpensive method for rapidly measuring the amount of drugs in EB.

If such a method becomes available it can be used by law enforcement and in doctors' offices, hospital emergency rooms, ambulances and other government agencies, military bases and companies seeking to screen employees for drug abuse. Vox Biomedical proposes to develop a method for quantitatively detecting the presence of drugs in EB by means of Differential Mobility Spectrometry (DMS) developed at Draper Laboratories. DMS is a robust, datarich, ultra-trace, chemical detection technology that has been proven for numerous applications including air quality cabin monitoring on the International Space Station (ISS), chemical warfare agent detection, explosives detection, and drinking water analysis. Recently Draper has applied this device to breath analysis for the detection of lung diseases.

A clinical study is currently underway and initial results are promising. This project involves transferring this technology developed by Draper for lung infection detection to the detection of psychoactive drugs in exhaled breath. Phase I of the proposed program will investigate the DMS signatures of cannabinoids in the laboratory and defining the device's limits of detection. A small pilot study will also be performed to demonstrate feasibility for using breath analysis as a proxy for the concentration of cannabinoids in the blood.

ELIGIBILITY:
Inclusion Criteria

* Capable of understanding and complying with the protocol
* In good physical and mental health (normal physical exam, ECG, blood and urine chemistries
* Absence of history or laboratory evidence of diabetes)
* Body Mass Index between 18-30,
* Inclusive Age 21-50 years (age will be verified by driver's license or other valid form of identification)
* Have a stable living situation with current postal address.

Exclusion criteria

* Meets criteria for current alcohol or substance use disorders (Past alcohol or substance use disorders greater than 3 years ago is acceptable)
* Concurrent diagnosis of Axis 1 disorder be maintained on an antipsychotic or antidepressant medication
* Taking prescription medications except certain short-term anti-fungal agents and some topical creams for dermal condition
* Heavy alcohol drinkers (greater than 15 drinks per week)
* Tobacco use greater than 5 cigarettes per day
* History of major head trauma resulting in cognitive impairment or history of seizure disorder
* Heavy caffeine use (greater than 500 mg on a regular daily basis)
* Has active hepatitis and/or aspartate aminotransferase (AST), alanine aminotransferase (ALT)> 3x the upper limit of normal
* For female participants, a positive pregnancy test.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult male and female volunteers
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Breath/cannabinoids concentrations | 1 year
  Quantitatively measuring cannabinoids in exhaled breath

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States